CLINICAL TRIAL: NCT05209763
Title: Standard vs Intensive Rehabilitation and Nutrition Regimen for Inpatients at the Intensive Care Unit
Brief Title: Standard vs Intensive Rehabilitation and Nutrition Regimen for Inpatients at the ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22/RVO-FNOs/2021
Record Dates: First submitted 2021-09-23; First posted 2022-01-27 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Nutrition Disorders
Keywords: Rehabilitation; Nutrition regimen; Intensive care; Internal medicine
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, 2x2 factorial design, angle centre interventional study with randomisation 1:1:1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard rehabilitation (Active Comparator): patient exercises with physiotherapists, staff assists with normal activities during the day, activation, and mobilization in and out of bed according to the patient's ability.
  Interventions: Procedure: More intensive rehabilitation
- More intensive rehabilitation (Experimental): * patient exercises with physiotherapists, staff assists with normal activities during the day, activation, and mobilization in and out of bed according to the patient's ability.
  * patient daily exercises using the rehabilitation device MOTOmed Letto 2 for a minimum of 5 days, maximum duration not limited, minimum duration of exercise 20 minuts once daily
  * exercise duration will be recorded daily and total time (in hours) at the end of the hospital stay
  Interventions: Procedure: More intensive rehabilitation
- Standard nutrition (Active Comparator): - nutrition determined by the attending physician according to recommendations for age, type of acute illness and comorbidities
  Interventions: Dietary Supplement: More intensive nutrition
- More intensive nutrition (Experimental): determined by the attending physician according to recommendations for age, type of acute illness and comorbidity
  - in addition, the patient will be administered hydroxymethylbutyrate at a dose of 3 g/day and in case of hypovitaminosis D and serum Ca concentration up to 3.0 mmol/l, vitamin D will be administered at a dose of 3000 IU/day for 5 days
  Interventions: Dietary Supplement: More intensive nutrition

INTERVENTIONS:
Procedure: More intensive rehabilitation — Patient exercises with physiotherapists, staff assists with normal activities during the day, activation, and mobilization in and out of bed according to the patient's ability.
  Arms: More intensive rehabilitation; Standard rehabilitation
Dietary Supplement: More intensive nutrition — in addition, the patient will be administered hydroxymethylbutyrate at a dose of 3 g/day - in case of ONS indication (oral nutrition support, formerly "sipping") in this form (Ensure advance plus 2 times a day), in case of non-indication or impossibility or intolerance of this form then in the form of a food supplement (Myotec HMB). The minimum total dose delivered is 12 g/5 days.
  * in case of hypovitaminosis D and serum Ca concentration up to 3.0 mmol/l, vitamin D will be administered at a dose of 3000 IU/day - cumulative 15000 IU/5 days (missing dose can be given at the end of the cycle in one dose)
  * inclusion of probiotics in standard doses
  Arms: More intensive nutrition; Standard nutrition

SUMMARY:
Older patients often suffer from multiple illnesses that require acute hospitalization. The goal of medical work is not only to save lives and heal acutely ill people but also to maintain physical fitness and self-sufficiency. In acutely hospitalized patients, the investigators often observe a decrease in muscle mass and strength, a deterioration in overall fitness with the need for long follow-up care, and sometimes permanent help with normal daily activities. An important part of the treatment of every acute patient is the emphasis on adequate nutrition and physical activity. The aim of this study is to determine the most appropriate intensity of exercise and diet that will be best for acute patients and will lead to the maintenance/improvement of physical fitness and thus shorten the length of hospitalization.

DETAILED DESCRIPTION:
The goal of daily medical work is not only to save lives and cure acutely ill patients but also to maintain quality of life, minimize the risk of complications, and, in the ever-growing population of geriatric patients, to maintain functional ability and self-sufficiency. Acute diseases of the internal type are almost always associated with catabolism leading to proteolysis and exacerbation of malnutrition. Patients are then often observed to have loss of muscle strength and muscle mass, deterioration of fitness, and in geriatric patients, who often have limited functional reserve and loss of self-sufficiency with the need for long follow-up care and sometimes permanent assistance with activities of daily living.

In addition to treating the disease itself, it is important to provide adequate nutrition and to maintain muscle strength and subsequent self-sufficiency by activating patients and providing optimally targeted physiotherapy. Studies demonstrating the effect of intensive rehabilitation are very heterogeneous and often performed on a relatively small number of subjects. Also, the results of these studies and their meta-analyses are inconclusive. It cannot be clearly stated based on the current scientific knowledge that intensive rehabilitation influences important endpoints such as in-hospital mortality, length of hospital stay, or the incidence of nosocomial infections. Early rehabilitation in acutely ill patients does influence muscle mass, but these effects are rather short-term.3 The effect of nutrition itself, or of individual nutrients (vitamin D, hydroxymethyl butyrate, etc.) is well known, and recommendations for nutrition have been developed based on this scientific knowledge. There is very limited evidence for the benefit of combining intensive rehabilitation and nutrition at the same time. The investigators know from available work that this intervention increases muscle mass and improves self-sufficiency.

A very important and still evolving area of medicine is the gut microbiome. The number of bacteria in our digestive tract is approximately the same as the number of cells in our entire body. Some authors speak of the gut microbiome as a separate organ. Intestinal bacteria and their products have a proven effect on the immune system locally and systemically and influence a variety of metabolic processes (insulin sensitivity, appetite, lipid metabolism and storage, oxidative stress, influence on inflammation, etc.). Today, it is possible to talk about the gut-muscle axis and know that the composition of the gut microbiome influences muscle tissue and, conversely, physical activity has been shown to have a benefit on the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* patient admitted to the Intensive Care Unit of the Department of Internal Medicine and Cardiology, University Hospital Ostrava, for an acute illness of an internal nature; patients admitted to another department of the hospital whose transfer to the above-mentioned ICU (intensive care unit) was carried out within 24 hours of the start of hospitalization may also be included
* assumption of a minimum length of hospital stay of 5 days
* ability to give informed consent
* the patient has both lower limbs
* the patient can receive fluids and liquid food orally

Exclusion Criteria:

* patient admitted from another health care facility where he/she has been admitted for more than 48 hours
* terminal stage of disease (tumor or non-tumor)
* patient with neuromuscular disease (polymyositis, etc.)
* severe chronic disease associated with severe maldigestion (e.g., patient on parenteral home nutrition)
* patient is fully immobile for a long time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay/hours | Through study completion, an average of 2 years
  To compare length of hospital stay (primary endpoint = length of hospital stay/hours) in four patient groups - standard RHB (rehabilitation) and standard nutritional care (SS-1), standard RHB + intensive nutritional care (SI-2), intensive RHB and standard nutritional care (IS-3) and intensive RHB + intensive nutritional care (II-4).

SECONDARY OUTCOMES:
Nosocomial infections during hospitalization. | Through study completion, an average of 2 years
  Incidence of nosocomial infection during hospitalization (Y/N).
Rehospitalization within 3 months after discharge. | Rehospitalization within 3 months of discharge of hospital.
  Rehospitalization within 3 months of discharge of hospital (Y/N).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ostrava, Ostrava, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tipping CJ, Harrold M, Holland A, Romero L, Nisbet T, Hodgson CL. The effects of active mobilisation and rehabilitation in ICU on mortality and function: a systematic review. Intensive Care Med. 2017 Feb;43(2):171-183. doi: 10.1007/s00134-016-4612-0. Epub 2016 Nov 18. PMID 27864615
- [Background] Morris PE, Berry MJ, Files DC, Thompson JC, Hauser J, Flores L, Dhar S, Chmelo E, Lovato J, Case LD, Bakhru RN, Sarwal A, Parry SM, Campbell P, Mote A, Winkelman C, Hite RD, Nicklas B, Chatterjee A, Young MP. Standardized Rehabilitation and Hospital Length of Stay Among Patients With Acute Respiratory Failure: A Randomized Clinical Trial. JAMA. 2016 Jun 28;315(24):2694-702. doi: 10.1001/jama.2016.7201. PMID 27367766
- [Background] Fuke R, Hifumi T, Kondo Y, Hatakeyama J, Takei T, Yamakawa K, Inoue S, Nishida O. Early rehabilitation to prevent postintensive care syndrome in patients with critical illness: a systematic review and meta-analysis. BMJ Open. 2018 May 5;8(5):e019998. doi: 10.1136/bmjopen-2017-019998. PMID 29730622
- [Background] Kou K, Momosaki R, Miyazaki S, Wakabayashi H, Shamoto H. Impact of Nutrition Therapy and Rehabilitation on Acute and Critical Illness: A Systematic Review. J UOEH. 2019;41(3):303-315. doi: 10.7888/juoeh.41.303. PMID 31548485
- [Background] Ticinesi A, Lauretani F, Tana C, Nouvenne A, Ridolo E, Meschi T. Exercise and immune system as modulators of intestinal microbiome: implications for the gut-muscle axis hypothesis. Exerc Immunol Rev. 2019;25:84-95. PMID 30753131
- [Background] Ticinesi A, Lauretani F, Milani C, Nouvenne A, Tana C, Del Rio D, Maggio M, Ventura M, Meschi T. Aging Gut Microbiota at the Cross-Road between Nutrition, Physical Frailty, and Sarcopenia: Is There a Gut-Muscle Axis? Nutrients. 2017 Nov 30;9(12):1303. doi: 10.3390/nu9121303. PMID 29189738
- [Background] Casati M, Ferri E, Azzolino D, Cesari M, Arosio B. Gut microbiota and physical frailty through the mediation of sarcopenia. Exp Gerontol. 2019 Sep;124:110639. doi: 10.1016/j.exger.2019.110639. Epub 2019 Jun 18. PMID 31226349